CLINICAL TRIAL: NCT00372476
Title: Open-label Trial of Imatinib in Combination With Vinorelbine for Patients With Advanced Breast Carcinoma: ICON
Brief Title: Efficacy and Safety of Imatinib and Vinorelbine in Patients With Advanced Breast Cancer
Acronym: INV181
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSTI571BDE28; 2005-001537-15
Record Dates: First submitted 2006-09-06; First posted 2006-09-07 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Tyrosine inhibitor; Chemotherapy; Imatinib
MeSH Terms: conditions — Breast Neoplasms | interventions — Imatinib Mesylate; Vinorelbine

ARMS (1):
- Imatinib + Vinorelbine (Experimental)
  Interventions: Drug: Imatinib and Vinorelbine

INTERVENTIONS:
Drug: Imatinib and Vinorelbine

SUMMARY:
This study is designed to investigate the safety and efficacy of the combination of imatinib and vinorelbine in patients with advanced, anthracycline resistant breast cancer

ELIGIBILITY:
Inclusion criteria:

* Histologically documented diagnosis of invasive breast cancer that is locally advanced or metastatic
* Previous anthracycline containing chemotherapy
* Presence of a certain protein on the cell surface (c-kit (CD117) and /or PDGF-receptor)
* Preferably tumor samples should be taken within 6 weeks of study entry. Most recent primary tumor tissue has to be available for analysis
* Acceptable health status (Eastern Cooperative Oncology Group [ECOG]-performance status 0,1, 2 or 3)

Exclusion criteria: (for the second-line therapy)

* Patient with Grade III/IV cardiac problems (i.e., congestive heart failure, myocardial infarction within 6 months of study) and with severe and/or uncontrolled medical disease (i.e., uncontrolled diabetes, chronic renal disease, or active uncontrolled infection).
* Patient has a known brain metastasis, chronic liver disease (i.e., chronic active hepatitis, and cirrhosis) and diagnosis of (HIV) infection.
* Patient received chemotherapy within 4 weeks prior to study entry, unless the disease is rapidly progressing.
* Patient previously received radiotherapy to ≥ 25 % of the bone marrow and had a major surgery within 2 weeks prior to study entry.
* Patient received either Vinorelbine or Imatinib in previous treatment regimens

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2006-06; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | at least 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Novartis Pharmaceuticals, Study Director — Novartis Pharmeceuticals
Locations (1):
- Novartis Investigative Site, Kiel, Germany

REFERENCES:
- [Result] Maass N, Schem C, Bauerschlag DO, Tiemann K, Schaefer FW, Hanson S, Muth M, Baier M, Weigel MT, Wenners AS, Alkatout I, Bauer M, Jonat W, Mundhenke C. Final safety and efficacy analysis of a phase I/II trial with imatinib and vinorelbine for patients with metastatic breast cancer. Oncology. 2014;87(5):300-10. doi: 10.1159/000365553. Epub 2014 Aug 26. PMID 25171229